CLINICAL TRIAL: NCT02880449
Title: Promoting Physical Activity Among Older Women Living in Socio-economically Disadvantaged Areas Using a Social Practice Theory Based Intervention: A Pilot Trial
Brief Title: Promoting Physical Activity Among Older Women Living in Socio-economically Disadvantaged Areas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Dr Mark Tully, Lecturer, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16.38
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Physical Activity; Health Behaviour
MeSH Terms: conditions — Motor Activity | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention will be conducted in pre-existing older women's groups based in community centres. The intervention will consist of three educational sessions, encouragement to enlist the support of a partner or 'buddy' (e.g. a spouse, partner or friend), an information pack (containing information on the local area, walking routes, points of interest) and the option of weekly telephone contact. Participants will be given the opportunity to discuss their progress and share feedback with the rest of the group at weekly meetings.
  Interventions: Behavioral: Intervention
- Control (No Intervention): Due to the stepped wedge design of the study, one group in each centre will not receive the intervention procedure detailed above until week seven. The control groups shall be given information about the study at baseline and informed that they will receive the intervention 6 weeks later.

INTERVENTIONS:
Behavioral: Intervention — A PA promoting intervention which provides education, social support and information about local opportunities for PA to pre-existing groups of older women living in socio-economically disadvantaged areas
  Arms: Intervention

SUMMARY:
The aim of the project is pilot an intervention to promote physical activity (PA) among older women.

Participants will be women aged ≥50 years attending an identified community centre situated in a socioeconomically deprived area of Belfast. The intervention consists of education, social support and information on local opportunities for physical activity (PA), based on Social Practice Theory. A stepped wedge design shall be used. The intervention was developed using findings from a literature review, systematic review and interviews with stakeholders. Outcome measures are accelerometer data, self-reported PA, a mental health questionnaire and qualitative interviews.

DETAILED DESCRIPTION:
Participants will be recruited from previously established older women's community groups. The intervention will utilize existing weekly community group sessions. A stepped wedge design, with a delayed intervention, shall be used to allow a randomised controlled trial to be conducted and to control for seasonal weather effects on PA levels. Two community groups from each centre shall be identified. One group from each centre shall receive the intervention from week one for 6 weeks; the second group shall receive the control condition from week one for 6 weeks and then receive the intervention at week 7 for 6 weeks. The intervention will consist of three educational sessions, encouragement to enlist the support of a partner or 'buddy' (e.g. a spouse, partner or friend), an information pack (containing information on the local area, walking routes, points of interest) and the option of weekly telephone contact. At each weekly meeting, participants will be given the opportunity to discuss their progress and share feedback with the rest of the group to gain peer social support. The intervention was developed using findings from a literature review, systematic review and interviews with stakeholders. The intervention is underpinned by constructs from the Social Practice Theory, a model that facilities behaviour change through the three elements of: materials (information on the local area, telephone calls, interactive group sessions), meanings (benefits of increasing PA, improving physical health and mental well-being) and competencies (encouragement to seek social support, knowledge of how to increase PA, knowledge of the local area).

ELIGIBILITY:
Inclusion Criteria:

* Females
* Aged over 50 years
* Member of women's community centres in an area of socioeconomic deprivation

Exclusion Criteria:

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Total number of steps per day | Baseline, 12 weeks and 6 months
  Changes from baseline number of steps per day measured objectively using an Actigraph accelerometer over a period of seven days.

SECONDARY OUTCOMES:
Mental health | Baseline, 12 weeks and 6 months
  To measure changes in mental health, using the HADS questionnaire, completed by participants
Moderate to vigorous physical activity (MVPA) | Baseline, 12 weeks and 6 months
  Changes from baseline in mean daily minutes of moderate physical activity (MVPA) measured objectively using an Actigraph accelerometer over a period of seven days.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Public Health, Queen's University Belfast, Belfast, United Kingdom

REFERENCES:
- [Derived] Lawlor ER, Cupples ME, Donnelly M, Tully MA. Promoting physical activity among community groups of older women in socio-economically disadvantaged areas: randomised feasibility study. Trials. 2019 Apr 25;20(1):234. doi: 10.1186/s13063-019-3312-9. PMID 31023329